CLINICAL TRIAL: NCT05314673
Title: Preoperative Intra-lesional Bevacizumab Injection in Primary Pterygium in Tunisian Patients: A Randomized Controlled Prospective Study
Brief Title: Preoperative Bevacizumab Injection in Primary Pterygium in Tunisian Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Fattouma Bourguiba (Other)
Responsible Party: Principal Investigator, Khairallah Moncef, Professor, University Hospital Fattouma Bourguiba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LR18SP09
Record Dates: First submitted 2022-02-28; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Pterygium
Keywords: pterygium; bevacizumab; recurrence; Vascularity; subconjunctival
MeSH Terms: conditions — Pterygium; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Preoperative intralesional injection of bevacizumab + pterygium excision+ autograft (Active Comparator): Patients receiving intralesional injection of 0.05 ml (1.25 mg) of Bevacizumab, one month before surgical treatment. Surgical treatment consisted of lesion excision and conjunctival autograft performed by a single trained surgeon.
  Interventions: Drug: Preoperative Intra-lesional Bevacizumab Injection in primary pterygium
- pterygium excision+ autograft (Active Comparator): Patients undergoing only pterygium surgical treatment.
  Interventions: Procedure: pterygium surgery without adjunctive therapy

INTERVENTIONS:
Drug: Preoperative Intra-lesional Bevacizumab Injection in primary pterygium — The surgical technique featured:
  subconjunctival anesthetic (lidocaine 2%) injection 5 mm from limbus; excision of the pterygium, starting from its head, followed by pterygium body removal; exposition of a triangular-shaped bare scleral bed (3-4 mm) conjunctival autograft stitched limbus to limbus with 10/0 vicryl suture Any intraoperative complication was noted and was treated accordingly. All patients received dexamethasone + tobramycin eye drops postoperatively 4 times a day in the 1st week. The eye drops were tapered over 4 weeks.
  Patients were examined 30 days before bevacizumab injection (D-30), before surgery (day 0: D0) and then at D7, M1, M3, and M6 after surgery.
  Arms: Preoperative intralesional injection of bevacizumab + pterygium excision+ autograft
Procedure: pterygium surgery without adjunctive therapy — The surgical technique featured:
  subconjunctival anesthetic (lidocaine 2%) injection 5 mm from limbus; excision of the pterygium, starting from its head, followed by pterygium body removal; exposition of a triangular-shaped bare scleral bed (3-4 mm) conjunctival autograft stitched limbus to limbus with 10/0 vicryl suture
  Arms: pterygium excision+ autograft

SUMMARY:
Purpose: To assess the efficacy and safety of a single preoperative intra-lesional bevacizumab injection in primary pterygium.

Methods: The investigators conducted a randomized controlled interventional study from January 2019 to December 2020. The study included a total of 60 patients (60 eyes) with primary pterygium. The investigators defined two groups of 30 patients each. Group A received an intralesional injection of bevacizumab (Avastin), one month before surgery (lesion excision and conjunctival autograft). Group B (control) had only the surgical treatment. Patients were followed up seven days (D7), one month (M1), three months (M3), and six months (M6) post-operatively. Pre-, per- and post-operatively, photographs of the lesions were taken, as well as a pathological examination. The main outcome measures were the change in functional discomfort following intralesional bevacizumab injection and pterygium recurrence. Recurrence was defined by fibrovascular tissue growth extending more than 1 mm across the limbus. Therapeutic success was defined as the absence of pterygium recurrence in M6.

DETAILED DESCRIPTION:
This prospective randomized controlled study adhered to the tenets of the Declaration of Helsinki. The Ethics Committee of our institution approved its modalities. The investigators had informed consent from all participants. The study included a total of 60 eyes of 60 patients with primary pterygium between January 2019 and December 2020. The investigators divided the patients into two groups of 30 patients each. The investigators performed a simple randomization method using a table of random numbers. Group A received an intralesional injection of 0.05 ml (1.25 mg) of Bevacizumab, one month before surgical treatment (lesion excision and conjunctival autograft by a single trained surgeon). Group B (control) had only the surgical treatment.

Each patient underwent a complete ocular examination: BSCVA, refraction, slit-lamp biomicroscopy, fundoscopy, and intraocular pressure measurement.

The investigators classified pterygium according to its stage (the Vaniscotte et al. Classification), grade (according to Tan et al. grading scheme), and color intensity (according to Teng et al : 0 = unremarkable, 1 = trace, 2 = mild, 3 = moderate, 4 = diffuse). The investigators measured Its corneal surface with Image J software. The study included patients over 18-years-old having primary pterygium with surgical indications:

* Stages 2, 3 and 4
* Significant astigmatism > 1.50 PD
* Patients with significant functional signs: according to a discomfort score that The investigators proposed.

Non-inclusion criteria were recurrent pterygium, suspected pterygium (sentinel vessels, resistant inflammation), and filtering surgery indication. Excluded were patients lost to follow-up or having a bevacizumab contraindication (hypertension, bleeding tendencies, previous myoredial infarction or stroke, pregnant and lactating women).

Pre-operative data gathered included basic demographic information (age and sex), medical and ophthalmological history, and involved eye(s).

The subjective variables: 1) photophobia; 2) foreign body sensation; 3) Ocular itching; 4) tearing, and 5) ocular redness; 6) visual blur, were evaluated according to their severity from 0 to 10 (visual analog scale (VAS)). The investigators assessed this score in each visit.

The surgical technique featured :

1. subconjunctival anesthetic (lidocaine 2%) injection 5 mm from limbus;
2. excision of the pterygium, starting from its head, followed by pterygium body removal;
3. exposition of a triangular-shaped bare scleral bed (3-4 mm)
4. conjunctival autograft stitched limbus to limbus with 10/0 vicryl suture Any intraoperative complication was noted and was treated accordingly. All cases were given dexamethasone + tobramycin eye drops postoperatively 4 times a day in the 1st week. The eye drops were tapered over 4 weeks.

Patients were examined 30 days before Bevacizumab injection (D-30) and surgery and then at D7, M1, M3, and M6 after surgery. The investigators assessed recurrence at each visit. Both groups (day 0: D0) had a per-operative histopathological examination.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of primary pterygium (stages 2,3 and 4) with surgical indication.

Exclusion Criteria:

* unable to attend the whole follow-up
* Bevacizumab contraindications (hypertension, bleeding tendencies, previous myocardial infarction or stroke, pregnant and lactating women).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of recurrence | 6 months post-operatively
  growth of fibrovascular tissue extending more than 1 mm across the limbus.
Rate of functional discomfort following intralesional bevacizumab injection | 6 months post-operatively
  The subjective variables: 1) photophobia; 2) foreign body sensation; 3) Ocular itching; 4) tearing; 5) ocular redness; and 6) visual blurring, were evaluated according to their severity from 0 to 10 (visual analogue scale (VAS)).

SECONDARY OUTCOMES:
Rate of mean changes from baseline in BCSVA | 6 months post-operatively
  one Snellen line
Rate of mean changes from baseline in astigmatism | 6 months post-operatively
  Astigmatism change > 0.25
% of patients with change in morphology of pterygium after injection | one month
  We classified pterygium according to its stage (the Vaniscotte et al. Classification), grade (according to Tan et al. grading scheme), and color intensity (according to Teng et al: 0 = unremarkable, 1 = trace, 2 = mild, 3 = moderate, 4 = diffuse).

CONTACTS AND LOCATIONS:
Overall Officials: Moncef Khairallah, Principal Investigator — Monastir University Hospital
Locations (1):
- Dhouha Gouider, Aryanah, Illinois, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: They are available